CLINICAL TRIAL: NCT05553678
Title: Effects of Midazolam on the Occurrence of Intraoperative Movement in Patients Undergoing Unruptured Intracranial Aneurysm Clipping Surgery: a Prospective Randomized Controlled Trial
Brief Title: The Effect of MDZ on Movement During UIA Clipping
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chang-Hoon Koo, Assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UIA-MDZ
Record Dates: First submitted 2022-09-18; First posted 2022-09-23 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Intraoperative Movement
MeSH Terms: interventions — Midazolam; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): Midazolam (0.03 mg/kg/30 min) will administered during UIA clipping through microscope.
  Interventions: Drug: Midazolam
- Control group (Placebo Comparator): Normal saline (0.03 ml/kg/30 min) will administered during UIA clipping through microscope.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Midazolam — Midazolam (0.03 mg/kg/30 min) will administered during UIA clipping through microscope.
  Arms: treatment group
Drug: Normal saline — Normal saline (0.03 mg/ml/30 min) will administered during UIA clipping through microscope.
  Arms: Control group

SUMMARY:
This study is a randomized, controlled, double-blinded, and parallel design study. A total 64 patients will be randomized to receive midazolam or normal saline during unruptured intracranial aneurysm clipping surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo elective unruptured intracranial aneurysm clipping surgery
* American Society of Anesthesiologists grade 1,2,3
* age > 18 year old

Exclusion Criteria:

* Refuse to participate to the study
* Body Mass Index < 18.5 kg/m2 or > 35 kg/m2
* Allergic history of benzodiazepine
* Pregnant

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Intraoperative movement | During microscopic surgery
  Incidence

SECONDARY OUTCOMES:
Motor evoked potential amplitude | immediately postoperative surgery
  amplitude
Motor evoked potential Latency | immediately postoperative surgery
  Latency
Duration of mechanical ventilation time | End of surgery to extubation time
  duration
Duration of ICU stay | From date of ICU admission until the date of first discharge from ICU, assessed up to 1 week
  duration of ICU stay, day
Satisfaction score for intraoperative environment | immediately postoperative surgery
  using 11-point score (0=worst dissatisfied, 10=very sattisfied)
Postoperative delirium | Postoperative 24 hour
  Incidence

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Hoon Koo, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No